CLINICAL TRIAL: NCT05454592
Title: Peer-Presented Versus Mental Health Service Provider-Presented Mental Health Outreach Programs for University Students: Randomized Controlled Trial
Brief Title: Peer-Presented Versus Mental Health Service Provider-Presented Mental Health Outreach Programs for University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Nancy Heath, Distinguished James McGill Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-11-031
Record Dates: First submitted 2022-07-04; First posted 2022-07-12 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Stress; Self Efficacy; Social Support; Social Connectedness; Mindfulness; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer-presented group (Experimental): The online outreach program focused on four key areas of mental health resilience-building: dealing with stress, decreasing self-criticism, improving self-care and help-seeking behaviours, and enhancing social connections and social support. Using videos, interactive infographics, guided audio recordings, and podcasts, students were provided with clear descriptions of each area of mental health resilience as well as a variety of evidence-based strategies specifically targeting one or more of these areas. A first video was sent to students describing the online program, its overall focus, and how to access the skills-based strategies on the website's interactive resource library. Two subsequent videos then were sent to (a) help students with problem-solving for common challenges to strategy practice, and (b) maintain long-term strategy practice habits. To assess differences in terms of preference for deliverer, this video series was delivered by undergraduate students (i.e., peers).
  Interventions: Behavioral: Stress and Coping Online Outreach Program
- Mental health service provider-presented group (Experimental): The program focused on four areas of mental health resilience-building: dealing with stress, decreasing self-criticism, improving self-care and help-seeking behaviours, and enhancing social connections and social support. Using videos, infographics, guided audio recordings, and podcasts, students were provided with clear descriptions of each area of mental health resilience as well as a variety of evidence-based strategies specifically targeting one or more of these areas. A first video was sent to students describing the online program, its overall focus, and how to access the skills-based strategies on the website's interactive resource library. Two subsequent videos were then sent to (a) help students with problem-solving for common challenges to strategy practice, and (b) maintain long-term strategy practice habits. To assess differences in terms of preference for deliverer, this video series was delivered by mental health service providers.
  Interventions: Behavioral: Stress and Coping Online Outreach Program
- Wait-list comparison group (No Intervention): Participants in the wait-list comparison group did not receive any intervention throughout the duration of the study. However, they were asked to fill out the same baseline, post, and follow-up surveys as all other participants.

INTERVENTIONS:
Behavioral: Stress and Coping Online Outreach Program — 3 videos and a resource library disseminated over the course of 9 weeks.
  Arms: Mental health service provider-presented group; Peer-presented group

SUMMARY:
The overarching goal of the present study was to evaluate a MHSP-presented versus peer-presented mental health resilience skills-building online video outreach program against a wait-list comparison group.

DETAILED DESCRIPTION:
Participants were recruited using a study flyer distributed to students in-person on campus and online through email listservs, social media platforms, and from an existing database of university students who participated in previous studies and agreed to be followed-up with. Given the self-paced nature of the program, a staggered recruitment approach was used wherein new participants completed the online baseline questionnaires between January 2020 until early March 2020.

Participants were randomly assigned to one of the three groups (MHSP-presented, peer-presented, or a wait-list comparison group), while counterbalancing the three groups based on gender and preference for seeking help from MHSPs or peers (i.e., using results from the General Help-seeking Questionnaire). Two weeks after the baseline questionnaire was sent, participants in the intervention groups received either the MHSP-presented video or the peer-presented video (video 1) depending on which group they were randomly assigned to, as well as a link for access to the resource library. The following two videos were sent two weeks apart. Participants were encouraged to access the resource library over the duration of the program and were reminded with each video link sent. All participants then received post (T2) and follow-up measures (T3) 6 and 10 weeks following the baseline completion respectively. Participants in the wait-list comparison group were only asked to complete evaluation measures at the three time points (they only received the videos and resource library at the end of the study). Following completion of the study, students received an e-mail with a personalized profile indicating their individual scores on various measures and all participants received full access to the program resources (videos and resource library).

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible for the study if they were between 18- 29 years of age, given the unique stressors associated with the developmental period of emerging adulthood (18-29 years old).
* Participants were required to have access to the internet (at least weekly) as the study was completed entirely online.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 274 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Change in Stress | Week 1, 6 & 10
  The Perceived Stress Scale (PSS) is a widely used self-report measure of individuals' perception of stress. This measure contains 10 items in which participants indicate their experience of stress on a 5-point Likert scale (0 = never to 4 = very often). Items were adapted to reflect experiences during the past week and include statements such as "In the past week, how often have you felt difficulties were piling up so high that you could not overcome them?" Ratings were averaged across items such that higher scores represented greater perceived stress. The PSS has good reliability (Cronbach's α = .89), construct validity, and predictive validity with reports of psychological and physical symptoms. In the present study, the PSS had good internal consistency with Cronbach's alphas at T1, T2, and T3 were .86, .82, and .85, respectively.

SECONDARY OUTCOMES:
Change in Coping Self-efficacy | Week 1, 6 & 10
  The Coping Self-Efficacy Scale (CSES) is a measure of one's confidence in effectively engaging in coping behaviors in the face of challenges. This measure contains 26 items in which participants indicate confidence in their coping strategies when it comes to handling challenges and stressors on an 11-point Likert scale (0 = cannot do at all to 10 = certain can do). The CSES states "When things aren't going well for you, or when you're having problems how confident or certain are you that you can do the following:" and include statements such as "find solutions to your most difficult problems" and "see things from the other person's point of view during a heated argument." Higher scores on the CSES represent higher coping-self efficacy. The CSES has good internal consistency (Cronbach's α = .91), and test-retest reliability. In the present study, the CSES had good internal consistency, with Cronbach's alphas at T1, T2, and T3 being .92, .93, and .94, respectively.
Change in Social Support | Week 1, 6 & 10
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item self-report questionnaire developed to assess the subjective perception of social support adequacy from family, friends, and significant others. Items are rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). Sample items include "There is a special person who is around when I am in need" and "My family really tries to help me." Higher scores on the MSPSS represent higher perception of social support. The MSPSS has good reliability (Cronbach's alpha ranging from .81 to .98) and has good convergent and construct validity In the present study, the MSPSS has a good internal consistency, with Cronbach's alphas at T1, T2, and T3 of .89, .91, and .92, respectively.
Change in Social Connectedness | Week 1, 6 & 10
  The Social Connectedness Scale Revised (SCS-R) is a 20-item self-report questionnaire that assesses emotional distance of the self from both friends and society, along with maintaining a sense of closeness. Items are rated on a 6-point Likert scale (1 = strongly disagree to 6 = strongly agree). Sample items include "I feel distant from people" and "I am able to relate to my peers." Higher scores on the SCS-R represent higher perception of social connectedness. The SCS-R has good internal reliability (Cronbach's α = .92) and has good convergent and discriminant validity. In the present study, the SCS-R had good internal consistency, with Cronbach's alphas at T1, T2, and T3 of .90, .89, and .91, respectively.
Change in Mindfulness | Week 1, 6 & 10
  The Mindful Attention Awareness Scale (MAAS) measures individuals' dispositional mindfulness (i.e., general tendency to be mindful) by assessing the frequency of mindful states over time. The MAAS consists of 15 items asking participants to report the frequency with which they have certain experiences on a 6-point scale (1 = almost always to 6 = almost never). Sample items include descriptions of experiences such as, "I find myself preoccupied with the future or the past" and "I find myself doing things without paying attention." Scores for this measure are such that higher scores indicate higher levels of mindfulness. The MAAS has demonstrated strong internal consistency (Cronbach's α = .89), as well as high test-retest reliability, convergent and discriminant validity. In the present study, the MAAS had good internal consistency, with Cronbach's alphas at T1, T2, and T3 of .80, .79, and .91, respectively.
Change in Quality of life | Week 1, 6 & 10
  The World Health Organization's Quality of Life Brief questionnaire is a 26-item measure assessing individuals' perception of their life quality within the following domains: physical health, psychological health, social relationships, and their environment. Participants are asked to rate items related to their experience of their own quality of life such on a 5-point Likert scale (1 = not at all to 5 = extreme amount). Sample items include "To what extent do you feel that physical pain prevents you from doing what you need to do?" and "How satisfied are you with the conditions of your living place?" The WHOQOL-BREF shows decent reliability (Cronbach's α values for physical health, psychological health, social relationships, and environmental health were .65, .77, .52 and .79, respectively) and good internal consistency.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The informed consent forms have been shared through the McGill repository which are open access to all individuals.
Supporting Information: ICF
Time Frame: Available as of September 2021
URL: https://escholarship.mcgill.ca/concern/theses/k0698d63k

REFERENCES:
- [Derived] Bastien L, Boke BN, Mettler J, Zito S, Di Genova L, Romano V, Lewis SP, Whitley R, Iyer SN, Heath NL. Peer-Presented Versus Mental Health Service Provider-Presented Mental Health Outreach Programs for University Students: Randomized Controlled Trial. JMIR Ment Health. 2022 Jul 22;9(7):e34168. doi: 10.2196/34168. PMID 35762935